CLINICAL TRIAL: NCT06888297
Title: European Certification of Interventions in Support of Second Victims (RESCUE)
Brief Title: RESCUE: European Certification for Second Victim Support
Status: Enrolling by invitation | Type: Observational
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira Solves, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Other Study IDs: RESCUE - IG19113
Record Dates: First submitted 2025-02-24; First posted 2025-03-21 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Second Victim Phenomenon; Occupational Stress; Healthcare Workforce Well-Being; Patient Safety; Healthcare Quality; Support Interventions
Keywords: Second Victim Phenomenon; Healthcare Professionals; Occupational Stress; Peer Support Programs; Psychological Support in Healthcare; Patient Safety; Healthcare Workforce Well-Being; Certification of Support Interventions
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- RESCUE-Support Interventions: Healthcare institutions participating in the certification process for structured second victim support interventions.
- RESCUE-Peer Supporters: Healthcare professionals receiving certification as peer supporters to assist colleagues experiencing the second victim phenomenon.

SUMMARY:
The "second victim" phenomenon affects healthcare professionals who experience highly stressful events in their daily practice, potentially compromising their well-being and patient safety. Despite the need for structured support interventions, many European institutions lack formal programs to address this issue.

The RESCUE project responds to this need, building on the previous work of the ERNST Consortium (COST Action 19113). Its objective is to develop and validate two certification systems: one for second victim support interventions and another for training healthcare professionals as peer supporters. A mixed-methods approach will be used, incorporating expert consensus techniques (e.g., Delphi study and consensus conferences) and pilot studies in healthcare institutions across multiple European countries.

The study aims to establish European certification standards for second victim support interventions, improving support for healthcare professionals, increasing resilience, and reducing the impact of adverse events on clinical performance.

DETAILED DESCRIPTION:
The RESCUE project (European Certification of Interventions in Support of Second Victims) aims to develop and validate two certification systems to improve support for healthcare professionals who experience the second victim phenomenon. This phenomenon occurs when healthcare workers are involved in stressful or traumatic clinical events, potentially affecting their well-being and patient safety. Despite its significant impact, many European institutions lack structured support interventions to address this issue.

Background and Rationale:

The ERNST Consortium (COST Action 19113) identified a critical gap in support interventions for second victims. Over four years of research, the consortium developed an intervention model structured into five stages: prevention, self-care, peer support, structured professional support, and structured clinical support. The RESCUE project builds upon this work to create a European-wide certification system for second victim support interventions and peer supporter training.

Study Objectives:

The primary objective of the study is to implement and validate two complementary certification systems:

RESCUE-Interventions: Certification for structured support interventions in healthcare institutions.

RESCUE-Peer Supporters: Certification for healthcare professionals trained to provide peer support.

These certification systems will be developed through expert consensus techniques (Delphi study, consensus conferences) and validated through pilot studies in multiple European healthcare institutions.

Methodology:

This is an observational, descriptive study using a mixed-methods approach. The study will be conducted in four phases:

Phase 1: Definition of certification standards through expert consensus and literature review.

Phase 2: Pilot application of the certification system in selected European institutions (Austria, Belgium, Portugal, and Spain).

Phase 3: Evaluation of certification effectiveness through qualitative and quantitative assessments.

Phase 4: Finalization and dissemination of the certification framework.

Expected Impact:

By establishing a standardized certification system, RESCUE seeks to ensure that healthcare professionals receive appropriate training and institutional support when dealing with adverse events. The project aims to increase resilience, improve patient safety, and integrate second victim interventions into European healthcare systems.

Funding and Ethical Considerations:

The study is funded by COST Innovators Grants (CIG), European Cooperation in Science & Technology (Grant ID IG19113) and has received approval from the Comité de Ética de la Investigación del Hospital Universitario San Juan de Alicante.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (e.g., physicians, nurses, midwives, clinical managers, patient safety officers).
* A minimum of 5 years of experience in healthcare-related fields such as clinical management, patient safety, quality assurance, or second victim support interventions.
* Employed in a healthcare institution or involved in second victim support initiatives at the time of the study.
* Willing to participate in peer support training, intervention certification, or evaluation processes related to the RESCUE project.
* Able to provide informed consent to participate in the study.

Exclusion Criteria:

* Non-healthcare professionals or individuals without experience in patient safety, clinical management, or second victim support.
* Less than 5 years of professional experience in relevant fields.
* Not affiliated with a healthcare institution or not involved in second victim support activities.
* Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthcare professionals from various disciplines, including physicians, nurses, midwives, clinical managers, patient safety officers, and other professionals involved in patient care and healthcare quality. Participants will be selected from European healthcare institutions implementing second victim support interventions.
  The study will include experts with at least 5 years of experience in healthcare-related fields, particularly in clinical management, quality assurance, and second victim support programs. The population will be drawn from hospitals, primary care centers, and social care institutions in multiple European countries, including Austria, Belgium, Portugal, and Spain.
  The study aims to develop and validate certification systems for second victim support interventions and peer supporter training, ensuring that healthcare institutions provide structured and evidence-based emotional support for affected professionals.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Development of Two Certification Systems for Second Victim Support Interventions and Peer Supporters | From study start (January 2025) to certification system finalization (May 2025).
  The study will assess the successful development and definition of certification standards for second victim support interventions (RESCUE-Interventions) and for healthcare professionals trained as peer supporters (RESCUE-Peer Supporters). The certification standards for second victim support interventions (RESCUE-Interventions) and peer supporters (RESCUE-Peer Supporters) will be developed using expert consensus methodologies, including Delphi studies and consensus conferences. Metric: Successful definition and agreement on certification criteria, with at least 85% consensus among experts in Delphi rounds and consensus meetings.
Relevance of the RESCUE Certification System | From the start of pilot studies (July 2025) to the end of data collection (October 2025).
  This measure will assess the perceived relevance of the RESCUE certification system for second victim support interventions and peer supporter training. The evaluation will be conducted through an ad hoc survey completed by healthcare professionals from the institutions participating in the field study.
  Metric: Percentage of healthcare professionals rating the certification system as "fairly relevant" or "highly relevant" on a 5-point Likert scale, based on responses to the relevant items in the 20-item survey. A minimum of 85% of positive responses ("fairly relevant" or "highly relevant") is required for the certification system to be considered relevant.
Feasibility of the RESCUE Certification System | From the start of the pilot studies (July 2025) to the end of data collection (October 2025).
  This measure will assess the perceived feasibility of implementing the RESCUE certification system in healthcare institutions. The evaluation will be conducted through an ad hoc survey completed by healthcare professionals from the institutions participating in the field study.
  Metric: Percentage of healthcare professionals rating the implementation of the certification system as "fairly feasible" or "highly feasible" on a 5-point Likert scale, based on responses to the relevant items in the 20-item survey. A minimum of 85% of positive responses ("fairly feasible" or "highly feasible") is required for the certification system to be considered feasible.
Acceptability of the RESCUE Certification System | From the start of pilot studies (July 2025) to the end of data collection (October 2025).
  This measure will assess the perceived acceptability of the RESCUE certification system among healthcare professionals. The evaluation will be conducted hrough an ad hoc survey completed by staff from the institutions participating in the field study.
  Metric: Percentage of healthcare professionals rating the certification system as "fairly acceptable" or "highly acceptable" on a 5-point Likert scale, based on responses to the relevant items in the 20-item survey. A minimum of 85% of positive responses ("fairly acceptable" or "highly acceptable") is required for the certification system to be considered acceptable.

SECONDARY OUTCOMES:
Perceived Scalability of the RESCUE Certification System in European Healthcare Institutions | From the start of the pilot phase (July 2024) to the end of study (October 2025).
  The perceived scalability and sustainability of the RESCUE certification system for implementation in other institutions and European countries will be assessed.
  Metric: Opinions of key stakeholders (institutional leaders, policymakers, and healthcare professionals) regarding the feasibility of the system, measured through structured interviews with qualitative analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, San Juan, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
Researchers affiliated with academic or healthcare institutions may request access to the dataset by submitting a formal request to the principal investigator. Approval will be granted based on ethical guidelines and compliance with data protection regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Supporting information may be available after study completion and publication of primary results, expected in Q1 2026
Access Criteria: Documents will be shared upon request with researchers affiliated with academic or healthcare institutions, subject to ethical approval and compliance with data protection regulations.
URL: https://cost-rescue.eu/

REFERENCES:
- [Background] Seys D, Panella M, Russotto S, Strametz R, Joaquin Mira J, Van Wilder A, Godderis L, Vanhaecht K. In search of an international multidimensional action plan for second victim support: a narrative review. BMC Health Serv Res. 2023 Jul 31;23(1):816. doi: 10.1186/s12913-023-09637-8. PMID 37525127
- [Background] Mira JJ, Matarredona V, Tella S, Sousa P, Ribeiro Neves V, Strametz R, Lopez-Pineda A. Unveiling the hidden struggle of healthcare students as second victims through a systematic review. BMC Med Educ. 2024 Apr 8;24(1):378. doi: 10.1186/s12909-024-05336-y. PMID 38589877
- [Background] Harkanen M, Pineda AL, Tella S, Mahat S, Panella M, Ratti M, Vanhaecht K, Strametz R, Carrillo I, Rafferty AM, Wu AW, Anttila VJ, Mira JJ. The impact of emotional support on healthcare workers and students coping with COVID-19, and other SARS-CoV pandemics - a mixed-methods systematic review. BMC Health Serv Res. 2023 Jul 13;23(1):751. doi: 10.1186/s12913-023-09744-6. PMID 37443003
- [Background] Guerra-Paiva S, Lobao MJ, Simoes DG, Fernandes J, Donato H, Carrillo I, Mira JJ, Sousa P. Key factors for effective implementation of healthcare workers support interventions after patient safety incidents in health organisations: a scoping review. BMJ Open. 2023 Dec 27;13(12):e078118. doi: 10.1136/bmjopen-2023-078118. PMID 38151271
- [Background] Guerra-Paiva S, Carrillo I, Mira J, Fernandes J, Strametz R, Gil-Hernandez E, Sousa P. Developing Core Indicators for Evaluating Second Victim Programs: An International Consensus Approach. Int J Public Health. 2024 Aug 30;69:1607428. doi: 10.3389/ijph.2024.1607428. eCollection 2024. PMID 39280904
- [Background] Gil-Hernandez E, Carrillo I, Tumelty ME, Srulovici E, Vanhaecht K, Wallis KA, Giraldo P, Astier-Pena MP, Panella M, Guerra-Paiva S, Buttigieg S, Seys D, Strametz R, Mora AU, Mira JJ. How different countries respond to adverse events whilst patients' rights are protected. Med Sci Law. 2024 Apr;64(2):96-112. doi: 10.1177/00258024231182369. Epub 2023 Jun 27. PMID 37365924
- [Background] Mira J, Carillo I, Tella S, Vanhaecht K, Panella M, Seys D, Ungureanu MI, Sousa P, Buttigieg SC, Vella-Bonanno P, Popovici G, Srulovici E, Guerra-Paiva S, Knezevic B, Lorenzo S, Lachman P, Ushiro S, Scott SD, Wu A, Strametz R. The European Researchers' Network Working on Second Victim (ERNST) Policy Statement on the Second Victim Phenomenon for Increasing Patient Safety. Public Health Rev. 2024 Sep 18;45:1607175. doi: 10.3389/phrs.2024.1607175. eCollection 2024. PMID 39360222
- [Background] Carrillo I, Tella S, Strametz R, Vanhaecht K, Panella M, Guerra-Paiva S, et al. Studies on the second victim phenomenon and other related topics in the pan-European environment: The experience of ERNST Consortium members. J Patient Saf Risk Manag. 2022;27(2):59-65. doi: 10.1177/25160435221076985
- [Derived] Mira JJ, Potura E, Schroder K, Panella M, Sousa P, Knezevic B, Tella S, Strametz R; RESCUE. Standardizing second victim support: development of the RESCUE certification framework for health care institutions. BMC Health Serv Res. 2025 Nov 27;25(1):1539. doi: 10.1186/s12913-025-13741-2. PMID 41310735
- See also: Official website of the RESCUE project, providing information on the study protocol, objectives, and implementation of second victim support interventions — https://cost-rescue.eu/